CLINICAL TRIAL: NCT06890871
Title: Radiotherapy Combined with Immunotherapy and Anti-angiogenic Therapy in Patients with Advanced HER2-negative Breast Cancer：a Single-arm, Exploratory Clinical Study
Brief Title: Radiotherapy with Immunotherapy and Anti-Angiogenic Therapy for Advanced HER2-Negative Breast Cancer: a Single-Arm Study
Status: Enrolling by invitation | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Zhongnan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023156
Record Dates: First submitted 2025-03-18; First posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer, Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Intervention Model Description: Radiotherapy combined with Immunotherapy and anti-angiogenic therapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- advanced HER2-negative breast cancer (Experimental)
  Interventions: Radiation: Intensity-modulated radiotherapy; Drug: Immunotherapy Therapy

INTERVENTIONS:
Radiation: Intensity-modulated radiotherapy — Radiotherapy With Immunotherapy and Anti-Angiogenic Therapy
Drug: Immunotherapy Therapy — Radiotherapy With Immunotherapy and Anti-Angiogenic Therapy

SUMMARY:
The treatment options for advanced HER2-negative breast cancer are limited. The single or combined drug therapy has a short remission time. Moreover, after multiple lines of treatment, patients are often in an awkward situation of "no more drugs available". And through literature research, it has been found that there is a synergistic effect between immunotherapy and anti-angiogenic therapy, as well as between radiotherapy and immunotherapy. This study will provide new approaches for the treatment of advanced HER2-negative breast cancer in the second-line setting, and offer new evidence-based medical evidence for patients with advanced HER2-negative breast cancer in the era of immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old, and willing to participate in this clinical study;

  * Pathologically diagnosed as invasive breast cancer; patients with breast cancer confirmed by imaging to have distant metastasis;

    * HER-2 negative (0/1+/2+ and FISH negative), and the pathological status of ER, PR and PD-L1 has been detected;

      * ECOG score 0-2; ⑤ ≥ 2 measurable lesions (according to RECIST 1.1.);

        * At least one metastatic lesion that can receive safe radiotherapy (excluding bone metastasis lesions);

          ⑦ Expected survival time > 3 months;

          ⑧ HER2-negative breast cancer that has relapsed or metastasized after receiving ≥ 2 lines of systemic treatment;

          ⑨ Good function of major organs, and laboratory test data meet the following standards: (1) Blood routine: Absolute neutrophil count ≥ 1.5 × 109/L (or greater than the lower limit of normal value in the laboratory of the research center), platelet count ≥ 100 × 109/L, hemoglobin ≥ 90 g/L; (2) Liver function: Serum total bilirubin ≤ 1.5 times the upper limit of normal value (ULN), AST and ALT ≤ 2.5 times ULN, if the patient has liver metastasis, this standard is ≤ 5 times ULN; (3) Renal function: CrCl ≥ 60 ml/min / 1.73 m2 (calculated according to the Cockcroft-Gault formula);

          ⑩ Female subjects with reproductive capacity, and male subjects whose partner has reproductive capacity, need to adopt one medically approved contraceptive measure (such as intrauterine device, contraceptive pills or condoms) during the study treatment period, and at least 6 months after the last treatment;

          ⑪ Voluntarily join this study, sign the informed consent form, have good compliance, and cooperate with follow-up.

Exclusion Criteria:

* Within 6 months prior to the first administration of the drug, there is a history of gastrointestinal perforation and/or fistula;

  * There is a history of uncontrollable pleural effusion, pericardial effusion or peritoneal effusion that requires repeated drainage;

    * There is a history of any allergy to any component of adalimumab;

      * Has received any of the following treatments:

        1. Within 4 weeks before the first administration of the study drug, has received any other investigational drug or the time from the last investigational drug administration is no more than 5 half-lives;
        2. Has been enrolled in another clinical study at the same time, unless it is an observational (non-interventional) clinical study or a follow-up of an interventional clinical study;
        3. Has received anti-tumor treatment (including radiotherapy, chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biological therapy or tumor embolization) within 2 weeks before the first administration of the study drug;
        4. Has received corticosteroids (more than 10mg of prednisone equivalent daily dose) within 2 weeks before the first administration of the study drug. Routine chemotherapy pre-treatment with hormones is allowed without dose adjustment. Other special circumstances need to be communicated with the investigator. In the absence of active autoimmune diseases, inhalation or local use of corticosteroids and doses >10mg/day of prednisone efficacy dose are allowed as an alternative for adrenal cortical hormones;
        5. Has received an anti-tumor vaccine or has received live vaccines within 4 weeks before the first administration of the study drug;
        6. Has undergone major surgery within 6 months or has had severe trauma;
        7. The lesion area has received high-dose radiation therapy;
        8. Has received PD1/PD-L1 treatment within 6 months;

           * The toxicity of previous anti-tumor treatment has not recovered to ≤CTCAE 5.0 grade 1 (except for alopecia);

             * Has contraindications to radiotherapy;

               * Has active autoimmune diseases, autoimmune disease history (such as interstitial pneumonia, colitis, hepatitis, pituitary inflammation, vasculitis, nephritis, hyperthyroidism, hypothyroidism, including but not limited to some diseases or syndromes); Excluding vitiligo or cured childhood asthma/allergy, adult patients without any intervention after adulthood; Using stable doses of thyroid replacement hormones for autoimmune-mediated hypothyroidism; Using stable doses of insulin for type I diabetes;

                 * Has a history of immunodeficiency, including positive HIV test, or has other acquired or congenital immune deficiency diseases, or has a history of organ transplantation and allogeneic bone marrow transplantation, or has active hepatitis (refer to HBV DNA test value over 500 IU/ml or 2500 copies/mL); ⑨ The subject has poorly controlled clinical symptoms or diseases of the cardiovascular system, including but not limited to: (1) NYHA grade II or above heart failure; (2) unstable angina pectoris; (3) having had a myocardial infarction within 1 year; (4) having clinical significance of supraventricular or ventricular arrhythmias that have not been controlled by clinical intervention or still not controlled after clinical intervention;

                   ⑩ Has had a serious infection within 4 weeks before the first administration of the study drug (CTCAE 5.0 > grade 2), such as severe pneumonia, sepsis, infection complications, etc. that require hospitalization treatment; Baseline chest imaging examination indicates active pulmonary inflammation, symptoms and signs of infection or need oral or intravenous antibiotic treatment within 2 weeks before the first administration of the study drug, except for preventive use of antibiotics;

                   ⑪ Has a history of interstitial lung disease (excluding radiation pneumonitis or non-infectious pneumonia history that has not been treated with hormone therapy);

                   ⑫ Has active pulmonary tuberculosis infection found through medical history or CT examination, or has a history of active pulmonary tuberculosis infection within 1 year before enrollment, or has a history of active pulmonary tuberculosis infection more than 1 year ago but has not received regular treatment; ⑬ Within the 5 years prior to the first use of the investigational drug, the subject was diagnosed with any other malignant tumor, except for those with low-risk metastasis and mortality risks (5-year survival rate > 90%), such as well-treated basal cell or squamous cell skin cancer or cervical carcinoma in situ, which are excluded;

                   ⑭ Pregnant or lactating women;

                   ⑮ According to the investigator's judgment, the subject has other factors that may force them to prematurely terminate the study, such as having other serious diseases (including mental disorders) that require combined treatment, severely abnormal laboratory test values, family or social factors that may affect the safety of the subject or the collection of trial data.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-08-08 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | If the therapeutic effect is CR or PR, the subjects must undergo confirmation no later than 3 weeks (21 days) after the first evaluation.
  The proportion of subjects whose BOR was rated as CR or PR according to the RECIST 1.1 standard

CONTACTS AND LOCATIONS:
Locations (1):
- #169, Donghu Road, Wuchang District, Wuhan, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No